CLINICAL TRIAL: NCT07211321
Title: Exploring the Relationship of Diets Inflammatory, Gut Microbiota, and Sarcopenia: A Cross-Sectional Study
Brief Title: Linking Diet, Inflammation, Gut Microbiota, and Sarcopenia: A Cross-Sectional Study
Status: Recruiting | Type: Observational
Sponsor: Jianhua Ma (Other)
Responsible Party: Sponsor-Investigator, Jianhua Ma, Lecturer, LanZhou University
Organization: LanZhou University (Other)
Other Study IDs: IRB23070101; No. 23JRRA1064 (Other Grant/Funding Number: Science and Technology Department of Gansu Province)
Record Dates: First submitted 2025-09-17; First posted 2025-10-07 (Actual); Last update posted 2025-10-07 (Actual); Status verified 2025-09

CONDITIONS: Sarcopenia
MeSH Terms: conditions — Sarcopenia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Faecal and whole blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- sarcopenia group and control group
  Interventions: Other: No Intervention: Observational Cohort

INTERVENTIONS:
Other: No Intervention: Observational Cohort — No Intervention

SUMMARY:
Based on the analysis of dietary characteristics, gut microbiota diversity, and composition, this study investigates the relationships between the dietary inflammatory potential, gut microbiota, and sarcopenia. Furthermore, it explores the mediating role of gut microbiota in the association between the dietary inflammatory index and the risk of sarcopenia. The findings are expected to provide insights into the mechanisms through which dietary inflammation influences the development and progression of sarcopenia, and to offer a basis for dietary and nutritional interventions aimed at preventing or managing this condition.

ELIGIBILITY:
Inclusion Criteria:

* Permanent residents of the community aged 60 years or older.
* Continuous residence duration in the community for more than 5 years.

Exclusion Criteria:

* Taking medications known to affect muscle function (e.g., corticosteroids, protein supplements, muscle enhancers).
* Requiring walking assistance or having severe cognitive impairment that would preclude successful completion of assessments including bioelectrical impedance analysis (BIA), gait speed measurement, and handgrip strength testing.
* Presence of a cardiac pacemaker, which contraindicates BIA measurement.
* Diagnosis of one or more chronic diseases that significantly limit dietary intake.

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This community-based cross-sectional study enrolled permanent residents aged 60 years or older who had been living in the community for more than 5 years.
Sampling Method: Probability Sample
Enrollment: 1220 (Estimated)
Dates: Start 2024-04-16 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
The prevalence of sarcopenia | Through study completion, an average of 1 year
  The diagnosis of sarcopenia is confirmed according to the AWGS 2019 criteria, which requires the assessment of muscle strength, physical performance, and muscle mass.
Change in absolute abundance of Faecalibacterium prausnitzii | Through study completion, an average of 1 year
  16S rRNA absolute quantification was used to detect the microbial composition of the fecal samples.
Dietary Characteristics | Through study completion, an average of 1 year
  Dietary data were collected using a food frequency questionnaire (FFQ) to analyze dietary patterns and nutrient intake.

CONTACTS AND LOCATIONS:
Locations (1):
- Lanzhou university, Lanzhou, Gansu, China

IPD SHARING:
Plan to Share IPD: No